CLINICAL TRIAL: NCT01495143
Title: Microdialysis of Paraspinal Muscle in Healthy Volunteers and Patients Underwent Posterior Lumbar Fusion Surgery
Brief Title: Surgical Stress Measured by Microdialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-07-012-RAS
Record Dates: First submitted 2009-12-29; First posted 2011-12-19 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Trauma
Keywords: Glucose; Lactate pyruvate ratio; Glycerol; Paraspinal muscle; Microdialysis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy group (Active Comparator): Eight healthy volunteers (five males and three females) with a body mass index of 23.8 and without chronic metabolic disease or low back pain. They are all non-smokers and non-medicated.
  Interventions: Procedure: Posterolateral lumbar fusion surgery
- Surgery group (Experimental): Two MD catheters is placed in the paraspinal muscle at the level of midpoint of incision bilaterally.
  A reference catheter is placed in the deltoid muscle.
  Interventions: Procedure: Posterolateral lumbar fusion surgery

INTERVENTIONS:
Procedure: Posterolateral lumbar fusion surgery — Two MD catheters with 1% lidocaine 1-2 ml are placed in the paraspinal muscle.
  Other Names: Lumbar diseases

SUMMARY:
Paraspinal muscle damage is inevitable during conventional posterior lumbar fusion surgery. Minimal invasive surgery is postulated to result in less muscle damage and better outcome. The aim of this study is to monitor metabolic changes of the paraspinal muscle and to evaluate paraspinal muscle damage during surgery using microdialysis (MD).

DETAILED DESCRIPTION:
Posterior approach is a common and important surgical procedure for various lumbar diseases. Owing to the anatomy, the damage of paraspinal muscle is inevitable during conventional posterior lumbar fusion surgery. Degeneration and malfunction of the paraspinal muscle might associate with pain and inferior postoperative clinical outcome.

ELIGIBILITY:
Inclusion criteria:

* patients who undergo conventional instrumented posterolateral lumbar fusion.

Exclusion criteria:

* previous fusion
* chronic metabolic disease
* tumor or metastasis
* postoperative surgical complications and complications during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The glycerol concentration | Two hours
  To study whether the glucerol concentration can be used to evaluate surgery related paraspinal muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Gang Ren, MD, PhD, Principal Investigator — Orthopaedic Division, North Denmark Region, Aalborg University Hospital, Denmark